CLINICAL TRIAL: NCT00532831
Title: Characterisation of Asthma in Obese Subjects. Relationships Between Asthma and Obesity, Potential Mechanisms by Which Obesity Can Contribute to Asthma and Modify Treatment Responses
Brief Title: Characterisation of Asthma in Obese Subjects
Status: Completed | Type: Observational
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Louis-Philippe Boulet, MD, FRCPC, FCCP, Laval University
Other Study IDs: HL-Phen-OB-1243
Record Dates: First submitted 2007-09-18; First posted 2007-09-20 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Asthma; Obesity
MeSH Terms: conditions — Asthma; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — serum plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Obese asthmatics: Obese subjects with asthma (on inhaled bd only)
- Non-obese asthmatics: Non-obese subjects with asthma(on inhaled bd only)

SUMMARY:
Our hypothesis:

Obese subjects with a physician's made diagnosis of asthma have a poorer asthma control than asthmatics with normal weight, less variability of peak expiratory flows (PEF) and bronchodilator response,increased induced sputum and systemic markers of inflammation and an increased prevalence of atopy.

Obese subjects have an increased incidence of co-morbidities such as rhinosinusitis, gastroesophageal reflux and sleep apnea syndrome.

This study aims to determine if, in comparison with asthmatics with a normal weight, paired for age and sex, obese subjects with asthma (all not using anti-inflammatory agents) show:

* A more uncontrolled asthma, increased health care use and poorer quality of life
* A reduced response to bronchodilators and diurnal variability of expiratory flows
* More marked airway inflammation and evidences of a systemic inflammatory response
* An increased prevalence of co-morbidities which can influence the report of respiratory symptoms or the severity of the disease, such as esophageal reflux symptoms, upper airway disease (rhinitis) and sleep apnea syndrome or other sleep disorder.

DETAILED DESCRIPTION:
Questionnaires on respiratory symptoms, health care use, quality of life, medication and asthma control will be administered and a thoracic examination performed.

Spirometry and bronchodilator response, blood tests for inflammatory parameters, pH measurements in exhaled air condensate and sputum induction will be performed. Peak expiratory flows will be measured and recorded on a diary card during one week.

On the second visit, measures of lung volumes and a methacholine challenge will be performed.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 and over.
* in good health apart from asthma or obesity as determined by history and physical examination (no other condition which could influence the proposed tests).
* All will be non smokers or ex- smokers for more than six months with a smoking history of no more than 10 pack- years (i.e., one pack per day or its equivalent for 10 years.)
* Subjects will have a physician's made diagnosis of asthma and have received a bronchodilator prescription in the last year.

Exclusion Criteria:

* Use of asthma medications other than bronchodilators
* Subjects who are, in the opinion of the investigator, mentally or legally
* incapacitated thus preventing informed consent from being obtained.
* Subjects having a co-existing illness that precludes them from the trial.
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects wiil be selected from the Hospital asthma primary care clinic and from advertisements in newspapers. Their will be offered to participate to the study
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2005-08; Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Airway response to methacholine | two weeks

SECONDARY OUTCOMES:
lung volumes | Two weeks

CONTACTS AND LOCATIONS:
Overall Officials: Louis-Philippe Boulet, MD, Principal Investigator — Hôpital Laval
Locations (1):
- Centre de Recherche, Hôpital Laval, Québec, Quebec, Canada

REFERENCES:
- [Derived] Lessard A, Turcotte H, Cormier Y, Boulet LP. Obesity and asthma: a specific phenotype? Chest. 2008 Aug;134(2):317-323. doi: 10.1378/chest.07-2959. Epub 2008 Jul 18. PMID 18641097